CLINICAL TRIAL: NCT02157597
Title: Randomized Trial of Near-infrared Spectroscopy to Guide Intraoperative and Intensive Care Management in Children's Heart Surgery Requiring Cardiopulmonary Bypass
Brief Title: NIRS Guidance Trail in Children's Heart Surgery
Acronym: NIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: American Society of Anesthesiologists (Other); International Anesthesia Research Society (IARS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-1677
Record Dates: First submitted 2012-11-15; First posted 2014-06-06 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (Active Comparator): The control patients will have open display of the NIRS monitor in the OR, but recording without display in the CICU, along with a request to the surgical and intensive teams to react to the data in their usual way. The disparity between the OR and CICU reflect the current opinions of the clinicians in these different environments regarding the necessity of NIRS monitoring within their sphere of practice.
  In this way, continuous recording of cerebral and somatic oximetry will be made in all patients. However for control patients the monitor display will be switched off in the CICU using a pre-programmed research mode, which permits both ongoing recording and also the display of technical error messages (such as inadvertent disconnections or probe displacement).
  Interventions: Other: Control
- NIRS based management (Experimental): The trial interventions of NIRS based management consists of provision to the cardiac surgical and intensive care teams of a protocol to guide their interpretation of cerebral and somatic NIRS monitoring and interventions to try in the event of monitored desaturation during the pre- and post-bypass periods (when the circulation is perfused by the beating of the native heart). The investigators believe that there is insufficient data to inform an evidence-based protocol for the bypass phase of surgery, particularly regarding the interpretation of NIRS data under conditions of hypothermia.
  Interventions: Other: NIRS based management

INTERVENTIONS:
Other: NIRS based management — 1. Check NIRS, mechanics, muscle relaxation, hemodynamics, ventilation, hematocrit, surgical repair
  2. Deepen anesthesia with volatile or intravenous agent.
  3. Consider Extra-Corporeal Membrane Oxygenation (ECMO).
  Arms: NIRS based management
Other: Control — During the Control Arm, the medical team completes all tasks as clinically necessary and in the best medical interest of the patient, without any input from the study procedures
  Arms: Control Arm

SUMMARY:
Heart surgery in young children involves some risks. This study looks at a new type of monitor that may reduce these risks. Near Infrared Reflectance Spectroscopy (NIRS) aims to measure if enough blood reaches vital organs in the body. The investigators goal is to see if this shows problems developing sooner than usual. The investigators do not know at this time if they can improve the blood supply to the vital organs. The investigators main aim is to see which responses work the best. The NIRS monitor is approved by the U.S. Food and Drug Administration (FDA).

The investigators will also follow the progress of recovery after surgery in the Cardiac Intensive Care Unit (CICU). This will find out if using the NIRS monitor improves the outcome for children.

DETAILED DESCRIPTION:
The NIRS monitor will record information from the patient until he/she has been in the CICU for about 24 hours. The monitoring consists of small sticky pads placed on the child's forehead and trunk. These work like the pulse oximeter (oxygen monitor) that has been used for for the child already, but have a more sensitive detector.

NIRS data will be recorded in the operating room and in the CICU for all babies in the study. The NIRS values can be seen by the surgical and anesthesia teams in the operating room for all babies in the study. Once the patient is in the CICU, the NIRS values will be visible to the CICU team only if he/she is assigned to the intervention group. If he/she is assigned to the control group the NIRS values will not be visible to the CICU team. Currently, use of the NIRS monitor is not standard care in the CICU.

For half of the children in the study (intervention group) the team will follow a carefully designed plan on how to react to any changes seen. For the other half of the children (control group) the team will respond to any changes seen according to their standard practice. For the control group NIRS monitoring will occur in the operating room but not in the CICU. By using two groups, the investigators can compare the NIRS recordings. In this way the investigators will find out if blood supply to the tissues is altered.

No standard monitoring or treatments will be withheld from the patient.

Some extra urine tests will be taken in the 24 hours following surgery. They will be taken from the catheter inserted into the patient's bladder, as is standard for all heart surgery. No genetic tests will be done.

The patient will have usual medical care following the 24 hours of the study. The investigators will use the hospital's electronic notes to collect further information. This will include medications, routine labs and vital signs. The investigators may also call the family 60 days after surgery with a few simple questions about the patient's current state of health.

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective or emergency heart surgery
* under 6 months of age
* operation requiring cardiopulmonary bypass
* complex operation, defined as RACH-1 score 3 to 6 inclusive

Exclusion Criteria:

* weight less than 2 kg
* prematurity defined as less than or equal to 36 weeks post-concepional age at tme of operation
* preoperative renal failure defined as serum creatinine greater than 132 mmol/l
* major non-cardiac congenital anomalies or preoperative non-cardiac disease
* operation or any of its components not classified in the RACHS-1 system
* receiving preoperative mechanical circulatory support
* presence of known intracranial hematomas or cerebral arteriovenous malformations
* reoperation if previously enrolled

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2011-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Cumulative time that NIRS is below threshold (from continuous electronic recording of NIRS data) | participants will be followed for the duration of surgery and during the first 24 hours postop in the CICU, an expected average of 35 hours.
  The investigators will assess effects of NIRS guidance in two ways. The primary outcome measure is the cumulative time (AUC) that rScO2 is below threshold (from continuous electronic recording of NIRS data). rScO2 will be taken as the mean of left and right forehead sensor readings. AUC will be calculated before and after CPB in the OR and during the first 24 hours postop in the CICU, and summed. Initial analyses of primary outcome to compare treatment groups will be undertaken on an intention-to-treat basis.

SECONDARY OUTCOMES:
Associated outcomes to heart surgery | participants will be followed for the duration of surgery and the CICU stay, an expected average of 3 weeks.
  Secondary outcomes include number and types of interventions, number and type of adverse events in the OR before and after CPB and in the CICU (e.g. cardiac arrest [need for chest compressions, defibrillation,ECMO],duration of pre-CPB and post-CPB, and NIRS complications [e.g. pressure injury]) recorded by a study coordinator.

CONTACTS AND LOCATIONS:
Overall Officials: Jayant Nick Pratap, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided